CLINICAL TRIAL: NCT04895631
Title: 18F-Fluorocholine Positron Emission Tomography (PET) for the Detection of Parathyroid Adenomas
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Hope (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-32553
Record Dates: First submitted 2021-05-13; First posted 2021-05-20 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Hyperparathyroidism, Primary
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — fluorocholine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fluorocholine PET Imaging (Experimental): Patients will undergo a single fluorocholine PET imaging study prior to surgery.
  Interventions: Drug: 18F-Fluorocholine; Procedure: Positron emission tomography (PET)

INTERVENTIONS:
Drug: 18F-Fluorocholine — One-time injection of 4-7 millicurie (mCi)
  Other Names: Fluorocholine
Procedure: Positron emission tomography (PET) — Imaging technique that uses radioactive substances known as radiotracers to visualize and measure changes in metabolic processes, and in other physiological activities
  Other Names: PET

SUMMARY:
This is a prospective single arm single center Phase III study evaluating the ability of 18F-fluorocholine to detect the location of parathyroid adenomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the performance (accuracy) of 18F-fluorocholine PET in the detection of hyperfunctioning parathyroid glands in surgical patients with biochemically proven primary hyperparathyroidism.

OUTLINE:

Participants will receive a single dose of 18F-Fluorocholine at the time the participant undergoes a single imaging study using 18F-fluorocholine. Study related procedures will end after the study visit. Participants who undergo subsequent parathyroidectomy, will have the results reviewed and compared to the results from the imaging study

ELIGIBILITY:
Inclusion Criteria:

* Age >= 13 years.
* Biochemically proven hyperparathyroidism and an indication for surgery.
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Current Pregnancy.
* Patients unlikely to comply with study procedures, restrictions and requirements and judged by the Investigator to be unsuitable for study participation.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with true-positives (sensitivity) of 18F-Fluorocholine PET using sestamibi imaging | Up to 1 year
  Sensitivity of 18F-fluorocholine PET for the detection of abnormal parathyroid adenomas confirmed by pathology as compared to sestamibi imaging. Location of parathyroid adenoma at imaging as read by three blinded readers, will be correlated to the location at surgery. True positive will be defined as an adenoma on imaging in the same location as seen at surgery. Sensitivity will be reported by individual reader.
Proportion of participants with true-positives (sensitivity) of 18F-Fluorocholine PET using predefined threshold | Up to 1 year
  Sensitivity of 18F-fluorocholine PET for the detection of abnormal parathyroid adenomas confirmed by pathology compared to a predefined threshold. Location of parathyroid adenoma at imaging as read by three blinded readers, will be correlated to the location at surgery. True positive will be defined as an adenoma on imaging in the same location as seen at surgery. Sensitivity will be reported by individual reader.

SECONDARY OUTCOMES:
Detection rate of 18F-fluorocholine PET | Up to 1 year
  The detection rate of 18F-fluorocholine PET in participants who have not undergone surgical resection will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No